CLINICAL TRIAL: NCT01481051
Title: PPL GLAU 12: A Phase 2 Dose Evaluation Study for the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: A Dose Evaluation Study for the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 12
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension (OH)
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Latanoprost-PPDS — Sustained delivery for 12 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and duration of the L-PPDS (latanoprost punctal plug delivery system) at different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* Diagnosis of bilateral open angle glaucoma or ocular hypertension
* Unmedicated IOP must be ≥22mm Hg

Exclusion Criteria:

* Any significant vision loss in the last year
* No contact lens use for the length of the study
* Abnormal eye lids, eye infection, or diseases to the eye
* Recent eye surgery
* Uncontrolled medication conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline | 12 weeks to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Cadden, Study Director — QLT Inc.
Locations (6):
- United States (6):
  - Sall Research Medical Center, Inc, Artesia, California
  - Wolstan & Goldberg Eye Associates, Los Angeles, California
  - West Coast Eye Care Associates, San Diego, California
  - Coastal Research Associates, LLC, Roswell, Georgia
  - R and R Eye Associates, San Antonio, Texas
  - Rocky Mountain Eye Care Associates, Salt Lake City, Utah